CLINICAL TRIAL: NCT04252703
Title: 'MInimalist' or 'MOre Complete' Strategies for Revascularization in Octogenarians Presenting With Non-ST-elevation Acute Coronary Syndromes: The MIMOSA Trial
Brief Title: 'MInimalist' or 'MOre Complete' Strategies for Revascularization in Octogenarians
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very slow recruitment - only 3 patients randomised and then COVID-19
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Francis Joshi, Principal Investigator, Interventional Cardiologist, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-18020388
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Multi Vessel Coronary Artery Disease; Ischemic Heart Disease; Acute Coronary Syndrome; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis
Keywords: ischemic heart disease; multivessel; octogenarians; acute coronary syndrome
MeSH Terms: conditions — Myocardial Ischemia; Acute Coronary Syndrome; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimalist (Active Comparator): The 'Minimalist' strategy is PCI treatment of the culprit lesion only. Other coronary stenoses are to be managed medically. It is recognized that there may be multiple culprit lesions in such patients, though there are no data on how frequently this might be expected. Operators may elect to treat multiple putative culprit lesions in this case.
  Interventions: Procedure: Percutaneous coronary intervention (PCI)
- More complete (Experimental): The 'More complete' strategy is PCI of the culprit lesion and fractional flow reserve (FFR)- or instantaneous wave-free ratio (iFR)-guided treatment of other angiographically significant (> 50% diameter) stenoses amenable to coronary stenting in vessels with reference diameters ≥2.5mm. Physiological assessment is strongly encouraged but not mandatory for lesions of ≥90% angiographic stenosis. PCI of chronic total occlusions will not be attempted as part of the study.
  Interventions: Procedure: Percutaneous coronary intervention (PCI)

INTERVENTIONS:
Procedure: Percutaneous coronary intervention (PCI) — Invasive cardiac catheterization, balloon angioplasty and intracoronary stenting.

SUMMARY:
Older patients with co-morbidity are increasingly represented in interventional cardiology practice. They have been historically excluded from studies regarding the optimal management of NSTEACS. Though there are associated risks with invasive treatment, such patients likely derive the greatest absolute benefit from PCI. Small, though highly selective, studies suggest a routine invasive strategy may reduce the risk of recurrent myocardial infarction.

The study aims to include, as far as possible, an 'all-comers' population of patients aged 80 and above to define the optimum amount of revascularization required to achieve good outcomes and satisfactory symptom relief for this challenging cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥80 years
* Non-ST-elevation acute coronary syndromes, defined as per guidelines:

  * Ischaemic chest pain or equivalent AND either
  * Electrocardiography with persistent or transient ST-depression and/or T-wave inversion OR
  * Biomarker positive for myocardial necrosis
* Multi-vessel coronary artery disease, defined as the presence of an angiographic >90% diameter or FFR-(<0.81) or iFR-(<0.90) positive stenoses(29) in a non-culprit vessel of reference diameter ≥2.5mm.

Exclusion Criteria:

* Inability to give written informed consent
* Resuscitation from cardiac arrest
* Life expectancy <12 months
* Cardiogenic shock
* Ventricular arrhythmias refractory to treatment at the time of randomization
* Coronary artery disease not amenable to PCI
* Heart Team decision for coronary bypass surgery
* Type 2 myocardial infarction(30) or alternative diagnoses such as tako-tsubo cardiomyopathy, as defined by the operator in light of the clinical picture at presentation
* Estimated glomerular filtration rate (eGFR) <20mL/min/m2 (by Cockcroft-Gault formula)
* Documented anaphylaxis induced by iodinated contrast media
* Documented allergies to either aspirin, clopidogrel, ticagrelor or oral anticoagulants
* Any condition that, in the opinion of the investigator, contraindicates anticoagulant therapy or would have an unacceptable risk of bleeding, such as, but not limited to, the following:

  * Active internal bleeding
  * Bleeding diastheses precluding treatment with dual antiplatelet therapy and/or oral anticoagulation
  * Platelet count <90,000/μL at screening
  * Previous intracranial haemorrhage
  * Clinically significant gastrointestinal bleeding within 12 months before randomization
  * Known significant liver disease (e.g. acute hepatitis, chronic active hepatitis, cirrhosis), or liver function test (LFT) abnormalities at screening (confirmed with repeat testing): alanine transaminase (ALT) >5 times the upper limit of normal or ALT >3 times the upper limit of normal plus total bilirubin >2 times the upper limit of normal
  * Major surgery, biopsy of a parenchymal organ, or serious trauma (including head trauma) within the past 30 days
* Any active non-cutaneous malignancy

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of a composite endpoint of all-cause death, recurrent myocardial infarction, urgent unplanned revascularization, TIMI major bleeding and/or stroke at 12 months. | 12 months
  Components of composite endpoint as defined below.

SECONDARY OUTCOMES:
Incidence of Cardiac death | 12 months
  defined as death due to suspected cardiac cause (myocardial infarction, low-output heart failure or fatal arrhythmia
Incidence of Myocardial infarction | 12 months
  Periprocedural myocardial infarction is defined as a CK-MB x 5 upper limit of normal (ULN) with ECG or angiographic evidence of ischaemia, or CK-MB x 10 ULN
Incidence of Urgent unplanned revascularization | 12 months
  (of the coronary arteries by either PCI or coronary bypass surgery)
Incidence of TIMI major and minor bleeding | 12 months
  defined as any symptomatic intracranial haemorrhage or clinically overt signs of haemorrhage (including imaging) associated with a drop in haemoglobin of ≥ 5g/dL. Minor bleeding is defined as any clinically overt sign of haemorrhage (including imaging) that is associated with a fall in haemoglobin concentration of 3 to ≤5 g/dL.
Incidence of Stroke | 12 months
  Defined as a clinically apparent neurological event lasting ≥24 hours verified by cerebral computed tomography (CT) or magnetic resonance imaging (MRI)
Incidence of contrast-induced nephropathy after PCI | 72 hours after PCI
  Defined as a 25% relative increase, or a 44μmol/L absolute increase in serum creatinine within 72 hours of contrast exposure in the absence of an alternative explanation)
Seattle Angina Questionnaire score | 12 months
  Performed at study entry and at 12 months follow-up
EQ-5D-5L quality of life assessment | 12 months
  Performed at study entry and at 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Engstrøm, MD, PhD, Principal Investigator — Rigshospitalet, Denmark; Francis Joshi, MD,PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Cardiology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No